CLINICAL TRIAL: NCT05073731
Title: Investigation of the Effects of the Synchronized Telerehabilitation-based Upper Extremity Training Program on Hand-arm Function, Pain, Fatigue, Quality of Life, and Participation in People With Multiple Sclerosis
Brief Title: Telerehabilitation-based Upper Extremity Training in People With Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/23-20
Record Dates: First submitted 2021-09-25; First posted 2021-10-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronized Telerehabilitation (Experimental): Physical activity training aiming to increase hand/arm function and fine motor function will be applied via videoconference for 8 weeks, 2 days a week, in 45-60 minute sessions.
  Interventions: Other: Telerehabilitation-based Upper Extremity Training
- Asynchronous Telerehabilitation (Active Comparator): Exercise videos and exercise tracking form will be sent.
  Interventions: Other: Telerehabilitation-based Upper Extremity Training

INTERVENTIONS:
Other: Telerehabilitation-based Upper Extremity Training — Telerehabilitation has been defined as "the delivery of rehabilitation services through information and communication technologies".
  Synchronized telerehabilitation provides the participant with advantages such as customized treatment, instant feedback, and a social environment such as face-to-face training.

SUMMARY:
In this studly, the effects of an 8-week telerehabilitation-based upper extremity training in persons with multiple sclerosis will be investigated.

DETAILED DESCRIPTION:
Multiple sclerosis is a chronic, progressive, and demyelinating disease of the central nervous system that affects more than 2.5 million people worldwide and is more common in young adults. The most common clinical signs and symptoms include motor dysfunction, fatigue, spasticity, cognitive impairment, chronic pain, depression, decreased quality of life, and bladder and bowel dysfunction.

66% of people with MS have impaired upper extremity function. As a result of the deterioration in upper extremity function, the performance of many daily living activities affects performance. In conclusion, there is a decrease in the functional independence of individuals, quality of life, and participation in activities in the community.

Telerehabilitation has been defined as "the delivery of rehabilitation services through information and communication technologies." Synchronized telerehabilitation provides the participant with advantages such as customized treatment, instant feedback, and a social environment such as face-to-face training. Telerehabilitation has proven to be a valuable modality for people with MS by increasing physical activity and reducing fatigue.

In terms of telerehabilitation-based upper extremity exercise training results, the MS population is deficient. Considering the importance of bilateral hand/arm function in daily life, this deficiency in the telerehabilitation-based training effect is eliminated.

For this reason, the results of this study, which will be created for the development of upper extremity telerehabilitation strategies in MS patients, will aim to improve the hand/arm function and fine motor skills of people with MS, aiming to increase the quality of life of individuals and to participate more actively in society.

Persons who followed by the outpatient Multiple Sclerosis Clinic of Dokuz Eylül University Hospital will participate in the study. A total of 30 participants will randomly be divided into 2 groups as synchronized telerehabilitation group and asynchronous telerehabilitation group.

A physiotherapist will give physical activity training aiming to increase hand/arm function and fine motor function to the Synchronized Telerehabilitation Treatment Group via videoconference for eight weeks, two days a week, in 45-60 minute sessions. Exercise videos and exercise tracking forms will be sent to the Asynchronous Telerehabilitation Treatment Group, the control group, with the exercise intensity and intensity equalized and their progression every two weeks. Assessments will done at baseline, after 8 weeks (post-treatment) and at 8 weeks (follow-up). Assessments will be done by assessors who are blinded to the group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Having a definitive diagnosis of MS according to the 2017 McDonald criteria
* Being over 18 years old
* Having answered yes to the question "Do you experience restriction in your hand-arm function and fine motor skills while performing your functional activities in daily life, and does this restriction limit your activities?"
* To have sufficient computer knowledge or to have a relative who can help in this regard to participate in the study for people with MS in the telerehabilitation group
* Having a computer and active internet connection at home for individuals with MS in the telerehabilitation group
* To be willing to participate in the study.

Exclusion Criteria:

* Having a neurological disease other than MS
* Having a relapse 30 days before or during the study
* Having an orthopedic problem that may affect the function of the upper extremity
* Cognitive disability at a level that hinders assessment and treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-28 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Change from Baseline at 8 weeks
  The Nine-Hole Peg Test measures finger dexterity.

SECONDARY OUTCOMES:
Expanded Disability Status Scale | Baseline
  Expanded Disability Status Scale is a method of quantifying disability in multiple sclerosis. The Expanded Disability Status Scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Jamar Hand Dynamometer | Change from Baseline at 8 weeks
  The Jamar Hand Dynamometer will be used to measure isometric force and peak strength.
Arm Function in Multiple Sclerosis Questionnaire | Change from Baseline at 8 weeks
  Arm Function in Multiple Sclerosis Questionnaire is a unidimensional 31-item questionnaire for measuring arm function in MS. The total sum score ranged from 31 to 186 and a high score indicates a low degree of arm function.
Preference-based Multiple Sclerosis Index | Change from Baseline at 8 weeks
  The Preference-based Multiple Sclerosis Index is a brief patient-reported outcome measure of health-related quality of life that consists of 5 items: walking, fatigue, mood, concentration, and roles and responsibilities. The scoring algorithm ranges from 0 (dead) to 1 (perfect health).
The Modified Fatigue Impact Scale - 5 | Change from Baseline at 8 weeks
  The MFIS-5 measures the impact of fatigue on cognitive, physical and psychosocial function-considered by some authors to be three important sub-scales-in patients with MS. Each item is scored between 0 and 4, and a low score indicates a low degree of fatigue.
Sensewear Armband | Change from Baseline at 8 weeks
  The SenseWear Armband (SWA; Bodymedia, Pittsburgh, Pennsylvania, USA) is a lightweight metabolic monitor will be used to estimate energy expenditure.
Global Perceived Effect Scale | At 8 weeks
  The global perceived effect (GPE) scale is a commonly used method for measuring patients' assessment of their condition. In different studies, different questions can be modified according to different levels and response styles. In our study, we will be asked the patient, "How do you find your hand/arm function compared to pre-rehabilitation?". They will be asked to choose one of the options "much improved, a little improved, no change, a little d e t e r i o r a t i o n, or much deterioration than before rehabilitation".
Impact of Participation and Autonomy Questionnaire | Change from Baseline at 8 weeks
  The IPAQ is a questionnaire that focuses on autonomy and participation of people with chronic conditions. The participation score ranges from 0-128, and experience of problems scores ranged from 0-16, with higher scores reflecting more restrictions in participation (less community participation) and/or more experience of problems.
Brief Pain Inventory-Short Form | Change from Baseline at 8 weeks
  The Brief Pain Inventory - Short Form (BPI-sf) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning on a 10 point scale. Higher scores reflecting more pain.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Ozakbas, MD, Study Director — MS Outpatient Clinic, Dokuz Eylul University Hospital
Locations (1):
- School of Physical Therapy and Rehabilitation, Dokuz Eylül University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided